CLINICAL TRIAL: NCT01560715
Title: Phase 2 Study Of Autologous Bone Marrow-Derived Stem Cells Transplantation For Retinitis Pigmentosa
Brief Title: Autologous Bone Marrow-Derived Stem Cells Transplantation For Retinitis Pigmentosa
Acronym: RETICELL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rubens Camargo Siqueira, MD,PhD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rubens Siqueira
Record Dates: First submitted 2012-03-19; First posted 2012-03-22 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis pigmentosa; stem cell; bone marrow; retinal dysprophy
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: Test group (Experimental): Retinitis pigmentosa patients with best-corrected visual acuity (BCVA) worse than 20/200 or visual field less than 20 degrees
  Interventions: Biological: intravitreal injection of autologous bone marrow stem cells

INTERVENTIONS:
Biological: intravitreal injection of autologous bone marrow stem cells — One intravitreal injection of a 0.1-ml cell suspension containing around 10x106 bone marrow mononuclear stem cells(BMMSC). All treatments were performed by a single retinal specialist using topical proparacaine drops under sterile conditions (eyelid speculum and povidone-iodine). Autologous BMMSC were injected into the vitreous cavity using a 27 gauge needle inserted through the inferotemporal pars plana 3.0 - 3.5 mm posterior to the limbus. After the injection, central retinal artery perfusion was confirmed with indirect ophthalmoscopy. Patients were instructed to instill one drop of 0.3% ciprofloxacin into the injected eye four times daily for 1 week after the procedure.
  Other Names: autologous bone marrow stem cells

SUMMARY:
The purpose of this study is to evaluate the short-term safety and efficacy of a single intravitreal injection of autologous bone marrow stem cells in patients with retinitis pigmentosa.

DETAILED DESCRIPTION:
A prospective phase II, nonrandomized open-label study of retinitis pigmentosa patients with best-corrected ETDRS visual acuity (BCVA) worse than 20/200. Standardized ophthalmic evaluation will be perform at baseline and at weeks 1, 4,12 and 24 (±1) following intravitreal injection of 10 x 106 bone marrow stem cells/ 0,1ml . Three measures will be used to evaluate the short-term safety of intravitreal of ABMDSC: 1) severe visual loss, defined as a drop in 15 letters on ETDRS visual acuity scale; 2) decrease in ERG response; 3) decrease in 5 square degrees on visual field; secondary safety outcomes : 1) increase in intra-ocular inflammation defined herein as anterior chamber cells and flare higher than 3+ for more than 1 month after injection according to a classification described elsewhere ; 2) decrease in CMT more than 50um; 3)genesis of abnormal tissues (teratomas) or tumors; 4) qualitative changes in retinal or choroidal perfusion, like macular nonperfusion. Secondary outcome measures will be used to evaluate the short-term efficiency of intravitreal of ABMDSC: 1) improvement in ERG response; 2) increase in visual field: 3) increase in CSMT > 50um and not related to macular edema; 4) increase > 5 letters on BCVA

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of retinitis pigmentosa logarithm of minimum angle of resolution (logMAR) BCVA of 1.0 (Snellen equivalent, 20/200) or worse
* visual Field less than 20 degreees

Exclusion Criteria:

* previous ocular surgery other than cataract
* presence of cataract or other media opacity that would influence ocular fundus documentation and adequate ERG and visual field evaluation
* other ophthalmic disease like glaucoma and uveitis
* previous history of blood disorders like leukemia
* known allergy to fluorescein or indocyanine green
* known coagulation abnormalities or current use of anticoagulative medication other than aspirin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
ETDRS Visual acuity change | Day 1 to Day 365

CONTACTS AND LOCATIONS:
Overall Officials: Rubens C Siqueira, MD,PhD, Principal Investigator — Sao Paulo University
Locations (1):
- Centro de Pesquisa Rubens Siqueira, São José do Rio Preto, São Paulo, Brazil

REFERENCES:
- [Background] Siqueira RC, Messias A, Voltarelli JC, Scott IU, Jorge R. Intravitreal injection of autologous bone marrow-derived mononuclear cells for hereditary retinal dystrophy: a phase I trial. Retina. 2011 Jun;31(6):1207-14. doi: 10.1097/IAE.0b013e3181f9c242. PMID 21293313
- [Background] Siqueira RC, Messias A, Messias K, Arcieri RS, Ruiz MA, Souza NF, Martins LC, Jorge R. Quality of life in patients with retinitis pigmentosa submitted to intravitreal use of bone marrow-derived stem cells (Reticell -clinical trial). Stem Cell Res Ther. 2015 Mar 14;6(1):29. doi: 10.1186/s13287-015-0020-6. PMID 25890251
- [Background] Siqueira RC. Stem cell therapy in retinal diseases? Rev Bras Hematol Hemoter. 2012;34(3):222-6. doi: 10.5581/1516-8484.20120054. No abstract available. PMID 23049424
- [Background] Siqueira RC, Messias A, Voltarelli JC, Messias K, Arcieri RS, Jorge R. Resolution of macular oedema associated with retinitis pigmentosa after intravitreal use of autologous BM-derived hematopoietic stem cell transplantation. Bone Marrow Transplant. 2013 Apr;48(4):612-3. doi: 10.1038/bmt.2012.185. Epub 2012 Sep 24. No abstract available. PMID 23000646